CLINICAL TRIAL: NCT00854386
Title: The Effect of Intraoperative Fluid Restriction on Postoperative Outcomes in Video-assisted Thoracic Surgery (VATS) for Lung Resection
Brief Title: Effect of Intraoperative Fluid Restriction on Postoperative Outcomes in Video-assisted Thoracic Surgery (VATS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof Idit Matot, director Anesthesiology and intensive care unit, Tel Aviv sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-IM-0502-CTIL
Record Dates: First submitted 2009-02-25; First posted 2009-03-03 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Acute Lung Injury (ALI); Acure Respiratory Distress Syndrome (ARDS); Sepsis
Keywords: fluid management; VATS; ALI; ARDS
MeSH Terms: conditions — Acute Lung Injury; Sepsis | interventions — Hospitals, High-Volume; Hospitals, Low-Volume

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): liberal fluid administration group
  Interventions: Drug: liberal fluid administration
- 2 (Experimental): Restrictive fluid administration group
  Interventions: Drug: restrictive fluid administration

INTERVENTIONS:
Drug: liberal fluid administration — patients in the liberal group (LG) will receive 8 ml/kg•hr of ringer lactate (RL) solution
  Other Names: liberal; standard; control; high volume
  Arms: 1
Drug: restrictive fluid administration — Patients in the restrictive group (RG) will receive 2 ml/kg•hr of Ringer Lactate (RL) solution throughout the intraoperative period
  Other Names: restrictive; experimental; low volume
  Arms: 2

SUMMARY:
The objective of this study is to compare the effects of two intraoperative fluid regimens - restrictive versus liberal (standard)- on postoperative outcomes (e.g. cardiopulmonary complications, morbidity, mortality and duration of hospitalization) in lung resections via Video-assisted thoracic surgery (VATS).

DETAILED DESCRIPTION:
Working hypothesis and aims:

The aim of this study is to investigate the effect of restrictive versus standard intraoperative fluid regimen on cardiopulmonary mordibity and mortality after VATS for lung resection. Our study hypothesis is that restrictive intraoperative fluid administration in patients undergoing VATS, will lead to better outcomes compared to a liberal fluid regimen.

Methods:

After obtaining informed consent, patients will be randomly assigned to one of two groups-liberal-protocol group (LG) or restricted-protocol group (RG). Anesthetic and surgical management will be performed similarly and according to standards for both groups, with one exception: patients in the RG group will receive 2 ml/kg•hr whereas patients in the RL group will receive 8 ml/kg•hr of Ringer Lactate (RL) solution throughout the intraoperative period. Hemodynamic changes during this period will be treated pharmacologically unless indicated otherwise. Blood loss, in both groups, will be replaced with RL solution in a 3:1 volume replacement, and blood and/or blood products will be transfused when required. Postoperatively, pain and fluid management will be standardized for both groups, according to departmental routines. Patient assessment will be performed by a blinded assessor. The primary endpoints of the study will combine: the incidence of post-operative complications (pulmonary, cardiovascular, others), re-intubations, and readmitions to the ICU during primary hospitalization; number of patients readmitted to the hospital within 30 days of surgery.

The secondary endpoints will include length of hospital stay, differences in hematocrit, urea, creatinine concentrations and oxygen saturation immediately postoperatively, in the first and third postoperative days and with discharge, and the number of patients receiving transfusion of blood and blood products; time to extubation, time to sit/stand/walk/eat/drink (recovery data).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old, with ASA I-III, undergoing elective VATS for lobectomy (of at least 2 segments), segmentectomy or pneumonectomy in the Sourasky Medical Center.

Exclusion Criteria:

* Patients with a history of chronic renal insufficiency (creatinine > 1.5 of normal value), congestive heart failure or hepatic dysfunction.

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary complications | 30 postoperative days

SECONDARY OUTCOMES:
Length of hospital stay | 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, Prof, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv Sourasky medical center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Background] Licker M, de Perrot M, Spiliopoulos A, Robert J, Diaper J, Chevalley C, Tschopp JM. Risk factors for acute lung injury after thoracic surgery for lung cancer. Anesth Analg. 2003 Dec;97(6):1558-1565. doi: 10.1213/01.ANE.0000087799.85495.8A. PMID 14633519
- [Background] Slinger PD. Acute lung injury after pulmonary resection: more pieces of the puzzle. Anesth Analg. 2003 Dec;97(6):1555-1557. doi: 10.1213/01.ANE.0000098363.76962.A2. No abstract available. PMID 14633517
- [Background] Arieff AI. Fatal postoperative pulmonary edema: pathogenesis and literature review. Chest. 1999 May;115(5):1371-7. doi: 10.1378/chest.115.5.1371. PMID 10334155
- [Background] Alam N, Park BJ, Wilton A, Seshan VE, Bains MS, Downey RJ, Flores RM, Rizk N, Rusch VW, Amar D. Incidence and risk factors for lung injury after lung cancer resection. Ann Thorac Surg. 2007 Oct;84(4):1085-91; discussion 1091. doi: 10.1016/j.athoracsur.2007.05.053. PMID 17888952
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Holte K, Klarskov B, Christensen DS, Lund C, Nielsen KG, Bie P, Kehlet H. Liberal versus restrictive fluid administration to improve recovery after laparoscopic cholecystectomy: a randomized, double-blind study. Ann Surg. 2004 Nov;240(5):892-9. doi: 10.1097/01.sla.0000143269.96649.3b. PMID 15492573
- [Background] Weissberg D, Schachner A. Video-assisted thoracic surgery--state of the art. Ann Ital Chir. 2000 Sep-Oct;71(5):539-43. PMID 11217470
- [Derived] Matot I, Dery E, Bulgov Y, Cohen B, Paz J, Nesher N. Fluid management during video-assisted thoracoscopic surgery for lung resection: a randomized, controlled trial of effects on urinary output and postoperative renal function. J Thorac Cardiovasc Surg. 2013 Aug;146(2):461-6. doi: 10.1016/j.jtcvs.2013.02.015. Epub 2013 Apr 1. PMID 23558303